CLINICAL TRIAL: NCT02852889
Title: Internal Jugular Vein Distensibility to Predict Fluid Responsiveness in Patients After Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2016-077
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Surgery
Keywords: internal jugular vein distensibility,haemodynamics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- fluid responders: Patients whose stroke volume index increase by >10% in response to a 500-ml fluid bolus was defined as fluid responders.
- fluid non-responders: Patients whose stroke volume index increase by <10% in response to a 500-ml fluid bolus was defined as fluid non-responders.

SUMMARY:
The purpose of the study was to verify the efficacy of using internal jugular vein (IJV) size and distensibility as an index of fluid responsiveness in mechanically ventilated patients after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* hypotension
* oliguria
* high lactate level

Exclusion Criteria:

* cardiac arrhythmia
* clinically relevant tricuspid or mitral regurgitation, clinically relevant right heart failure
* thrombosis in any large upper body veins
* bilaterally inserted venous catheters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
fluid responsiveness （mean artery pressure、cardiac output、stroke volume variation、internal jugular vein distensibility） | after fluid challenge (30min)
  CO increased more than 10% was defined as fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Guo-wei Tu, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No